CLINICAL TRIAL: NCT02702414
Title: A Phase 2 Study of Pembrolizumab (MK-3475) as Monotherapy in Subjects With Advanced Hepatocellular Carcinoma (KEYNOTE-224)
Brief Title: Study of Pembrolizumab (MK-3475) as Monotherapy in Participants With Advanced Hepatocellular Carcinoma (MK-3475-224/KEYNOTE-224)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-224; MK-3475-224 (Other: MSD); KEYNOTE-224 (Other: MSD); 163434 (Other: JAPIC-CTI); 2015-004566-28 (EudraCT Number)
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Programmed Cell Death 1 (PD1, PD-1); Programmed Cell Death Ligand 1 (PDL1, PD-L1); Programmed Cell Death Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Hepatocellular Carcinoma (HCC)-Prior Systemic Therapy with Sorafenib (Experimental): Participants with previously systemically treated HCC received a pembrolizumab 200 mg intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations. Participants who stopped pembrolizumab as a result of obtaining a confirmed complete response (CR) or those who stopped after receiving 35 trial treatments were eligible for an additional 17 trial treatments (approximately an additional 1 year of treatment) after progressive disease if they met the criteria for re-treatment.
  Interventions: Biological: Pembrolizumab
- Cohort 2: HCC-Systemic Therapy Naïve (Experimental): Participants with HCC who had not received treatment for systemic disease received a pembrolizumab 200 mg IV infusion on Day 1 of each 3-week cycle for up to 35 administrations. Participants who stopped pembrolizumab as a result of obtaining a confirmed complete response (CR) or those who stopped after receiving 35 trial treatments were eligible for an additional 17 trial treatments (approximately an additional 1 year of treatment) after progressive disease if they met the criteria for re-treatment.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Intravenous (IV) infusion
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
This is a efficacy and safety study of pembrolizumab (MK-3475, KEYTRUDA®) as monotherapy in participants with hepatocellular carcinoma (HCC) in two cohorts: participants with advanced HCC and with no curative option after disease progression on sorafenib or intolerance of sorafenib (Cohort 1) or who had not received treatment for systemic disease (Cohort 2). Study participants may receive pembrolizumab once every 3 weeks for up to 35 initial cycles (up to approximately 2 years) and a potential additional 17 cycles in a re-treatment phase (approximately an additional 1 year of treatment) .

The primary objective of this study is to determine the Objective Response Rate (ORR) of pembrolizumab given as monotherapy in participants with HCC.

Effective with Amendment 7: Upon study completion, participants are discontinued and may be enrolled in a pembrolizumab extension study, if available.

ELIGIBILITY:
Inclusion Criteria:

* For Cohort 1: has histologically or cytologically confirmed diagnosis of HCC (fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible) based on pathology report
* For Cohort 2: has an HCC diagnosis confirmed by radiology, histology, or cytology (fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible)
* Has Barcelona Clinic Liver Cancer (BCLC) Stage C disease or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach
* Has a Child-Pugh Class A liver score within 7 days of first dose of study drug
* Has a predicted life expectancy >3 months
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as confirmed by the blinded central imaging vendor
* Has a performance status of 0 or 1 using the Eastern Cooperative Oncology Group (ECOG) Performance Scale within 7 days of first dose of study drug
* For Cohort 1: has documented objective radiographic progression after stopping treatment with sorafenib or else intolerance to sorafenib
* Is willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug (male and female participants of childbearing potential)
* Demonstrates adequate organ function

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy, herbal/complementary oral or intravenous (IV) medicine, or used an investigational device within 4 weeks of the first dose of study drug. Participant must also have recovered from associated therapy (i.e., to Grade ≤1 or baseline) and from adverse events due to any prior therapy
* For Cohort 1: has received sorafenib within 14 days of first dose of study drug
* Has had esophageal or gastric variceal bleeding within the last 6 months
* Has clinically apparent ascites on physical examination
* Has portal vein invasion at the main portal (Vp4), inferior vena cava, or cardiac involvement of HCC based on imaging
* Has had encephalopathy in the last 6 months. Participants on rifaximin or lactulose to control their encephalopathy are not allowed
* Had a solid organ or hematologic transplant
* For Cohort 1: had prior systemic therapy for HCC other than sorafenib, or intercurrent local therapy to the liver tumor between sorafenib and study drug
* For Cohort 2: had prior systemic therapy in the advanced disease setting
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs)
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has a diagnosed additional malignancy within 5 years for Cohort 1 and 3 years for Cohort 2 prior to first dose of study treatment with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected in situ cervical and/or breast cancers
* Has radiographically detectable central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has evidence or history of interstitial lung disease or active noninfectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a known severe hypersensitivity to pembrolizumab, its active substance and/or any of its excipients
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
* Has received prior immunotherapy including anti-programmed death-1 (anti-PD-1), anti-PD-ligand-1 (anti-PD-L1), or anti-PD-L2 agents, or if the participant has previously participated in clinical studies with pembrolizumab (MK-3475)
* Has a known history of human immunodeficiency virus (HIV)
* Has untreated active Hepatitis B virus (HBV)
* For Cohort 1: has dual infection with HBV/Hepatitis C virus (HCV) or other hepatitis combinations at study entry
* For Cohort 2: has dual active HBV infection (Hepatitis B surface antigen positive and/or detectable HBV deoxyribonucleic acid [DNA]) and HCV infection (detectable HCV ribonucleic acid [RNA]) at study entry
* Has received a live vaccine within 30 days of planned start of study drug (Cycle 1, Day 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Chan SL, Finn RS, Edeline J, Ogasawara S, Knox JJ, Daniele B, Ryoo BY, Merle P, Bouattour M, Lim HY, Chao Y, Yau T, Haber BA, Malhotra U, Siegel AB, Liu CC, Kudo M, Cheng AL. Effect of pembrolizumab on viral hepatitis load and transaminases in advanced hepatocellular carcinoma. Ann Hepatol. 2025 Dec 24;31(1):102169. doi: 10.1016/j.aohep.2025.102169. Online ahead of print. PMID 41453647
- [Derived] Zhou X, Cao J, Topatana W, Xie T, Chen T, Hu J, Li S, Juengpanic S, Lu Z, Zhang B, Wang K, Feng X, Shen J, Chen M. Evaluation of PD-L1 as a biomarker for immunotherapy for hepatocellular carcinoma: systematic review and meta-analysis. Immunotherapy. 2023 Apr;15(5):353-365. doi: 10.2217/imt-2022-0168. Epub 2023 Feb 27. PMID 36852452
- [Derived] Verset G, Borbath I, Karwal M, Verslype C, Van Vlierberghe H, Kardosh A, Zagonel V, Stal P, Sarker D, Palmer DH, Vogel A, Edeline J, Cattan S, Kudo M, Cheng AL, Ogasawara S, Daniele B, Chan SL, Knox JJ, Qin S, Siegel AB, Chisamore M, Hatogai K, Wang A, Finn RS, Zhu AX. Pembrolizumab Monotherapy for Previously Untreated Advanced Hepatocellular Carcinoma: Data from the Open-Label, Phase II KEYNOTE-224 Trial. Clin Cancer Res. 2022 Jun 13;28(12):2547-2554. doi: 10.1158/1078-0432.CCR-21-3807. PMID 35421228
- [Derived] Kudo M, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer DH, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Yau T, Gurary EB, Siegel AB, Wang A, Cheng AL, Zhu AX; KEYNOTE-224 Investigators. Updated efficacy and safety of KEYNOTE-224: a phase II study of pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib. Eur J Cancer. 2022 May;167:1-12. doi: 10.1016/j.ejca.2022.02.009. Epub 2022 Mar 29. PMID 35364421
- [Derived] Zhu AX, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer D, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Webber AL, Ebbinghaus SW, Ma J, Siegel AB, Cheng AL, Kudo M; KEYNOTE-224 investigators. Pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib (KEYNOTE-224): a non-randomised, open-label phase 2 trial. Lancet Oncol. 2018 Jul;19(7):940-952. doi: 10.1016/S1470-2045(18)30351-6. Epub 2018 Jun 3. PMID 29875066
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had 2 cohorts with each cohort starting treatment at a different time period during the study.
  One participant allocated to Cohort 1 withdrew from the study before receiving treatment. This participant was not eligible for safety or efficacy analysis.
Pre-assignment Details: Per protocol, final analyses of all outcome measures were planned to be performed during the first course of therapy and collection of adverse events and all-cause mortality were planned to be done in both first and second courses.
Period: Overall Study
Arm/Group | Cohort 1: Hepatocellular Carcinoma (HCC)-Prior Systemic Therapy With Sorafenib | Cohort 2: HCC-Systemic Therapy Naïve
Started | 105 | 51
Treated | 104 | 51
Received Second Course of Pembrolizumab | 4 | 1
Completed | 0 | 0
Not Completed | 105 | 51
Not completed — Death | 96 | 42
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Sponsor Decision | 8 | 7

BASELINE CHARACTERISTICS:
Population: All allocated participants
Groups:
- Cohort 1: HCC-Prior Systemic Therapy With Sorafenib: Participants with previously systemically treated HCC received a pembrolizumab 200 mg IV infusion on Day 1 of each 3-week cycle for up to 35 administrations. Participants who stopped pembrolizumab as a result of obtaining a confirmed complete response (CR) or those who stopped after receiving 35 trial treatments were eligible for an additional 17 trial treatments (approximately an additional 1 year of treatment) after progressive disease if they met the criteria for re-treatment.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: HCC-Prior Systemic Therapy With Sorafenib | Cohort 2: HCC-Systemic Therapy Naïve | Total
Number analyzed (Participants) | 105 | 51 | 156
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.4 (8.2) | 67.7 (10.3) | 67.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 7 | 26
  Male | 86 | 44 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 99 | 45 | 144
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 2 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 1 | 4
  White | 85 | 48 | 133
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a confirmed Complete Response (CR: Disappearance of all target and non-target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target and non-target lesions) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by blinded central imaging vendor. Participants with missing data were considered non-responders. The percentage of participants who experienced a CR or PR per RECIST 1.1 is presented.
Time Frame: Up to approximately 34 months for Cohort 1 and up to approximately 28 months for Cohort 2
Population: All participants who received at least one dose of study treatment during the first course of therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: HCC-Prior Systemic Therapy With Sorafenib | Cohort 2: HCC-Systemic Therapy Naïve
Number analyzed (Participants) | 104 | 51
Percentage of participants | 18.3 [11.4 to 27.1] | 15.7 [7.0 to 28.6]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR was determined in participants who demonstrated a confirmed Complete Response (CR: disappearance of all target and non-target lesions) or Partial Response (PR: ≥30% decrease in the sum of diameters of target and non-target lesions) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by blinded central imaging vendor. DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. Participants who had not progressed, started a new anti-cancer therapy, been lost to follow-up, or died at the time of analysis were censored at the date of their last tumor assessment. Per RECIST 1.1, PD was at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm, OR unequivocal progression for non-target lesions, OR appearance of one or more new lesions. The DOR per RECIST 1.1 for all participants who had a confirmed CR or PR is presented.
Time Frame: Up to approximately 34 months for Cohort 1 and up to approximately 28 months for Cohort 2
Population: All participants who received at least one dose of study treatment and who had a confirmed CR or confirmed PR during the first course of therapy.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: HCC-Prior Systemic Therapy With Sorafenib | Cohort 2: HCC-Systemic Therapy Naïve
Number analyzed (Participants) | 19 | 8
Months | 21.0 [10.7 to NA] — NA=upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse | 16.2 [3.1 to NA] — NA=upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who had a CR (disappearance of all target and non-target lesions), PR (at least a 30% decrease in the sum of diameters of target and non-target lesions), or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD was at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm, OR unequivocal progression for non-target lesions, OR appearance of one or more new lesions.]). CR, PR, and SD were evaluated per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by blinded central imaging vendor. Participants with missing data were considered as participants whose disease was not under control. The percentage of participants who experienced a confirmed CR, PR, or SD is reported.
Time Frame: Up to approximately 34 months for Cohort 1 and up to approximately 28 months for Cohort 2
Population: All participants who received at least one dose of study treatment during the first course of therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: HCC-Prior Systemic Therapy With Sorafenib | Cohort 2: HCC-Systemic Therapy Naïve
Number analyzed (Participants) | 104 | 51
Percentage of participants | 61.5 [51.5 to 70.9] | 56.9 [42.2 to 70.7]

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from the first dose to the first documented disease progression per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by blinded central imaging vendor. PD was at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm, OR unequivocal progression for non-target lesions, OR appearance of one or more new lesions. If there was no documented disease progression, TTP was censored at last tumor assessment date. The TTP was analyzed using the product-limit (Kaplan-Meier) method for censored data. TTP per RECIST 1.1 is presented.
Time Frame: Up to approximately 34 months for Cohort 1 and up to approximately 28 months for Cohort 2
Population: All participants who received at least one dose of study treatment during the first course of therapy.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: HCC-Prior Systemic Therapy With Sorafenib | Cohort 2: HCC-Systemic Therapy Naïve
Number analyzed (Participants) | 104 | 51
Months | 4.8 [3.9 to 7.0] | 4.4 [2.5 to 8.6]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the first dose to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by blinded central imaging vendor. PD was at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm, OR unequivocal progression for non-target lesions, OR appearance of one or more new lesions. If there was no disease progression or death, participants were censored at the date of their last disease assessment. The PFS was analyzed using the product-limit (Kaplan-Meier) method for censored data. PFS is presented.
Time Frame: Up to approximately 34 months for Cohort 1 and up to approximately 28 months for Cohort 2
Population: All participants who received at least one dose of study treatment during the first course of therapy.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: HCC-Prior Systemic Therapy With Sorafenib | Cohort 2: HCC-Systemic Therapy Naïve
Number analyzed (Participants) | 104 | 51
Months | 4.9 [3.5 to 6.7] | 4.3 [2.1 to 7.8]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was determined for all participants and was defined as the time from the first dose to death due to any cause. Participants were censored at the last known alive date. The OS was analyzed using the product-limit (Kaplan-Meier) method for censored data. The OS is presented.
Time Frame: Up to approximately 34 months for Cohort 1 and up to approximately 28 months for Cohort 2
Population: All participants who received at least one dose of study treatment during the first course of therapy.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: HCC-Prior Systemic Therapy With Sorafenib | Cohort 2: HCC-Systemic Therapy Naïve
Number analyzed (Participants) | 104 | 51
Months | 13.2 [9.7 to 15.3] | 16.9 [8.3 to 23.1]

7. Secondary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. The number of participants who experienced at least one AE is presented. Per protocol, final analysis for this outcome measure was planned to be performed during the first course of therapy only.
Time Frame: Up to approximately 34 months for Cohort 1 and up to approximately 28 months for Cohort 2
Population: All participants who received at least one dose of study treatment during the first course of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HCC-Prior Systemic Therapy With Sorafenib | Cohort 2: HCC-Systemic Therapy Naïve
Number analyzed (Participants) | 104 | 51
Participants | 101 | 49

8. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. The number of participants who discontinued study treatment due to an AE is presented. Per protocol, final analysis for this outcome measure was planned to be performed during the first course of therapy only.
Time Frame: Up to approximately 34 months for Cohort 1 and up to approximately 28 months for Cohort 2
Population: All participants who received at least one dose of study treatment during the first course of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HCC-Prior Systemic Therapy With Sorafenib | Cohort 2: HCC-Systemic Therapy Naïve
Number analyzed (Participants) | 104 | 51
Participants | 23 | 8

ADVERSE EVENTS:
Time Frame: Up to approximately 87 months
Description: All-cause mortality (ACM)=all allocated participants; AEs=all participants who received ≥1 dose of treatment. Per protocol, disease progression was not considered an AE unless related to treatment. Medical Dictionary for Regulatory Activities (MedDRA) terms neoplasm progression (NP), malignant NP, and disease progression not related to treatment were excluded. Per protocol, collection of AEs and ACM were planned for both first and second courses and reported separately.
Groups:
- Cohort 1: Hepatocellular Carcinoma (HCC)-Prior Systemic Therapy With Sorafenib-First Course: Participants with previously systemically treated HCC received a pembrolizumab 200 mg IV infusion on Day 1 of each 3-week cycle for up to 35 administrations. Participants who stopped pembrolizumab as a result of obtaining a confirmed complete response (CR) or those who stopped after receiving 35 trial treatments were eligible for an additional 17 trial treatments (approximately an additional 1 year of treatment) after progressive disease if they met the criteria for re-treatment.
- Cohort 2: HCC-Systemic Therapy Naïve-First Course: Participants with HCC who had not received treatment for systemic disease received a pembrolizumab 200 mg IV infusion on Day 1 of each 3-week cycle for up to 35 administrations. Participants who stopped pembrolizumab as a result of obtaining a confirmed complete response (CR) or those who stopped after receiving 35 trial treatments were eligible for an additional 17 trial treatments (approximately an additional 1 year of treatment) after progressive disease if they met the criteria for re-treatment.
- Cohort 1: Hepatocellular Carcinoma (HCC)-Prior Systemic Therapy With Sorafenib-Second Course: Participants from Cohort 1 who met the criteria for re-treatment received a pembrolizumab 200 mg IV infusion on Day 1 of each 3-week cycle for up to 17 administrations.
- Cohort 2: HCC-Systemic Therapy Naïve-Second Course: Participants from Cohort 2 who met the criteria for re-treatment received a pembrolizumab 200 mg IV infusion on Day 1 of each 3-week cycle for up to 17 administrations.
Arm/Group | Cohort 1: Hepatocellular Carcinoma (HCC)-Prior Systemic Therapy With Sorafenib-First Course | Cohort 2: HCC-Systemic Therapy Naïve-First Course | Cohort 1: Hepatocellular Carcinoma (HCC)-Prior Systemic Therapy With Sorafenib-Second Course | Cohort 2: HCC-Systemic Therapy Naïve-Second Course
All-Cause Mortality (participants affected / at risk) | 94/105 | 42/51 | 2/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 44/104 | 21/51 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 96/104 | 46/51 | 4/4 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Hepatocellular Carcinoma (HCC)-Prior Systemic Therapy With Sorafenib-First Course (N=104) | Cohort 2: HCC-Systemic Therapy Naïve-First Course (N=51) | Cohort 1: Hepatocellular Carcinoma (HCC)-Prior Systemic Therapy With Sorafenib-Second Course (N=4) | Cohort 2: HCC-Systemic Therapy Naïve-Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Hepatocellular Carcinoma (HCC)-Prior Systemic Therapy With Sorafenib-First Course (N=104) | Cohort 2: HCC-Systemic Therapy Naïve-First Course (N=51) | Cohort 1: Hepatocellular Carcinoma (HCC)-Prior Systemic Therapy With Sorafenib-Second Course (N=4) | Cohort 2: HCC-Systemic Therapy Naïve-Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 11 (12) | 1 (1) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 8 (9) | 6 (6) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 16 (18) | 8 (9) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 10 (13) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 12 (12) | 6 (6) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 18 (18) | 4 (4) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 17 (21) | 13 (15) | 1 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 21 (21) | 4 (6) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (15) | 3 (3) | 0 (0) | 0 (0)
Asthenia (General disorders) | 16 (19) | 7 (8) | 1 (1) | 0 (0)
Fatigue (General disorders) | 30 (40) | 21 (23) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (3) | 3 (4) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 20 (21) | 14 (15) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 5 (6) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (4) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 13 (16) | 3 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 23 (27) | 3 (3) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 6 (7) | 2 (2) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 9 (10) | 3 (3) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 16 (18) | 8 (9) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (31) | 5 (8) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (16) | 5 (6) | 2 (4) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (10) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 4 (4) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 8 (10) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 6 (6) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 24 (29) | 6 (8) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 14 (19) | 5 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT02702414/Prot_SAP_001.pdf